CLINICAL TRIAL: NCT06695117
Title: A Phase 1/2, Parallel, Randomized, Modified Double-blind, Multi-arm Study to Assess the Safety and Immunogenicity of a Combination Vaccine Comprised of Different Recombinant Spike Antigen Levels of a Matrix-M Adjuvanted Recombinant COVID-19 Vaccine and High-dose Inactivated Influenza Vaccine in Adult Participants 50 Years of Age and Older
Brief Title: Study of a Combination Vaccine Comprised of Different Recombinant Spike Antigen Levels of a Matrix-M Adjuvanted Recombinant COVID-19 Vaccine and High-Dose Inactivated Influenza Vaccine in Adult Participants 50 Years of Age and Older
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VBT00001; U1111-1310-5034 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Immunization; Influenza Immunization
Keywords: COVID-19 Vaccine and Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be performed in a modified double-blind fashion.
  Modified double-blind:
  * Investigator, participants, and laboratory personnel will be blinded
  * Clinical site staff preparing/administering the study vaccines will be unblinded
  * Sponsor study staff will be blinded, except for dedicated staff involved in interim analysis, who will be unblinded at the time of interim analysis, and for dedicated staff involved in assessing criteria for safety surveillance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1: IIV-HD (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: IIV-HD; Other: Placebo (0.9% NaCl)
- Group 2: rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: rC19 (dose 1); Other: Placebo (0.9% NaCl)
- Group 3: IIV-HD (in right or left deltoid) and rC19 (dose1) (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: IIV-HD; Biological: rC19 (dose 1)
- Group 4: IIV-HD + rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: IIV-HD + rC19 (dose 1); Other: Placebo (0.9% NaCl)
- Group 5: IIV-HD + rC19 (dose 2) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: IIV-HD + rC19 (dose 2); Other: Placebo (0.9% NaCl)
- Group 6: IIV-HD + rC19 (dose 3) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: IIV-HD + rC19 (dose 3); Other: Placebo (0.9% NaCl)
- Group 7: IIV-HD + rC19 (dose 4) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: IIV-HD + rC19 (dose 4); Other: Placebo (0.9% NaCl)

INTERVENTIONS:
Biological: IIV-HD — Inactivated, split-virion
  Arms: Group 1: IIV-HD (in right or left deltoid) and placebo (in opposite deltoid); Group 3: IIV-HD (in right or left deltoid) and rC19 (dose1) (in opposite deltoid)
Biological: rC19 (dose 1) — Protein subunit
  Arms: Group 2: rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid); Group 3: IIV-HD (in right or left deltoid) and rC19 (dose1) (in opposite deltoid)
Biological: IIV-HD + rC19 (dose 1) — IIV-HD component: Inactivated, split-virion rC19 component: Protein subunit
  Arms: Group 4: IIV-HD + rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid)
Biological: IIV-HD + rC19 (dose 2) — IIV-HD component: Inactivated, split-virion rC19 component: Protein subunit
  Arms: Group 5: IIV-HD + rC19 (dose 2) (in right or left deltoid) and placebo (in opposite deltoid)
Biological: IIV-HD + rC19 (dose 3) — IIV-HD component: Inactivated, split-virion rC19 component: Protein subunit
  Arms: Group 6: IIV-HD + rC19 (dose 3) (in right or left deltoid) and placebo (in opposite deltoid)
Biological: IIV-HD + rC19 (dose 4) — IIV-HD component: Inactivated, split-virion rC19 component: Protein subunit
  Arms: Group 7: IIV-HD + rC19 (dose 4) (in right or left deltoid) and placebo (in opposite deltoid)
Other: Placebo (0.9% NaCl) — Normal saline
  Arms: Group 1: IIV-HD (in right or left deltoid) and placebo (in opposite deltoid); Group 2: rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid); Group 4: IIV-HD + rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid); Group 5: IIV-HD + rC19 (dose 2) (in right or left deltoid) and placebo (in opposite deltoid); Group 6: IIV-HD + rC19 (dose 3) (in right or left deltoid) and placebo (in opposite deltoid); Group 7: IIV-HD + rC19 (dose 4) (in right or left deltoid) and placebo (in opposite deltoid)

SUMMARY:
Study VBT00001 is planned to be a Phase 1/2, randomized, modified double-blind, active-controlled, multi-center study to be conducted in approximately 980 adults aged 50 years and older in the United States.

The purpose of the study is to assess the safety and immunogenicity of IIV-HD (high-dose inactivated influenza vaccine) + rC19 (adjuvanted recombinant COVID-19 vaccine) vaccine comprised of IIV-HD combined with different recombinant Spike (rS) antigen levels of rC19 compared to IIV-HD alone, rC19 (dose 1) alone, and IIV-HD and rC19 (dose 1) (coadministered in opposite arms).

Placebo will be coadministered in the IIV-HD alone, rC19 (dose 1) alone, and IIV-HD + rC19 study groups to control for the number of injections and to maintain observer-blinding.

Thus, each participant will receive two injections at enrollment, one in each deltoid muscle.

Study details include:

* The study duration will be approximately 12 months
* Study intervention will be administered via a single intramuscular (IM) injection into the right and left deltoid muscles on D01
* Dose escalation with sequential enrollment (sentinel cohort followed by main cohort for a given dose)
* The visit frequency will be D01, D09 (telephone call), D30, D182 (telephone call), and D366 (telephone call)

Number of Participants:

Approximately 980 participants are expected to be randomized.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria to be checked at Screening Visit

* Aged 50 years or older on the day of inclusion
* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all study procedures.
* Participant must be able to receive an injection in the deltoid muscle of both arms.
* Participant must have completed a primary vaccination series against SARS-CoV-2 and at least 1 booster with a locally authorized or approved COVID-19 vaccine.

Inclusion criteria to be checked at Visit 1 (D01):

* Aged 50 years or older on the day of inclusion
* Participants who are healthy or with pre-existing stable condition (defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 12 weeks before enrollment), as determined by medical evaluation including medical history and physical examination.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.

OR

• Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration.

A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) on the day of enrollment before the first dose of study intervention.

* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all study procedures.
* Participant must be able to receive an injection in the deltoid muscle of both arms.
* Participant must have completed a primary vaccination series against SARS-CoV-2 and at least 1 booster with a locally authorized or approved COVID-19 vaccine.

Exclusion Criteria:

Exclusion criteria to be checked at Screening Visit and at Visit 1 (D01):

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (for glucocorticoids, ≥ 10 milligrams/day of prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances .
* Self-reported thrombocytopenia, contraindicating intramuscular injection, based on investigator's judgment.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection, based on investigator's judgment.
* Chronic illness (1) that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion .
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 100.4°F) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* History of serious adverse reaction to any influenza or COVID-19 vaccines.
* Personal or family history of Guillain-Barré syndrome.
* Prior history of myocarditis, pericarditis, or myopericarditis.
* Prior history of stroke, transient ischemic attack, or stroke risk factors, which may include untreated/uncontrolled hypertension, untreated/uncontrolled hyperlipidemia, active smoking, atrial fibrillation, and additional risk factors, based on investigator's judgment, which may include history of thromboembolic disease, obesity, cardiac structural or valvular abnormality, carotid stent placement, or family history of stroke..
* Receipt of any vaccine in the 4 weeks preceding study intervention administration or planned receipt of any vaccine prior to the second blood draw (ie, approximately in the 28 days following study intervention administration .
* Previous vaccination against influenza (in the previous 6 months) with an investigational or marketed vaccine.
* Previous vaccination against COVID-19 (in the previous 6 months) with an investigational or marketed vaccine OR history of COVID-19 in the previous 6 months .
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Participation at the time of study enrollment (or in the 4 weeks preceding study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Deprived of freedom by an administrative or court order, or being in an emergency setting, or hospitalized involuntarily.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

  1. Chronic illness may include, but is not limited to, cardiac disorders, hypertension, pulmonary disease, renal disorders, auto-immune disorders, diabetes mellitus, psychiatric disorders, neurologic disorders, or chronic infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Within 30 minutes after each vaccination
  Immediate adverse events are any unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site reactions | Up to 7 each days after vaccination
  Solicited injection site reactions include injection site pain, erythema and swelling
Number of participants with solicited systemic reactions | Up to 7 days after each vaccination
  Solicited systemic reactions include fever, headache, fatigue, myalgia and chills
Number of participants with unsolicited AEs | Up to 28 days after each vaccination
  Unsolicited (spontaneously reported) AEs, not fulfilling criteria for solicited adverse reactions
Number of participants with adverse events of special interest (AESIs) | Up to 180 days after each vaccination
  AESIs
Number of participants with medical attended adverse events (MAAEs) | Up to 180 days after each vaccination
  MAAEs
Number of MAAEs relating to predefined potential immune-mediated disease (PIMDs) | From D182 through 12 months following the last study vaccination
  MAAEs relating to predefined PIMDs
Number of participants with serious adverse events (SAEs) | Up to 180 days after each vaccination
  SAEs
Number of participants with related SAEs | From D182 through 12 months following the last study vaccination
  Related SAEs
Number of MAAEs relating to predefined PIMDs that meet the criteria for SAEs | From D182 through 12 months following the last study vaccination
  MAAEs relating to predefined PIMDs that meet the criteria for SAEs
Geometric mean (GM) of HAI titers in all participants | At D01 and D30
  HAI titers
Geometric mean ratio (GMR) HAI titers ratio D30/D01 in all participants | At D01 and D30
  Individual HAI titers ratio D30/D01
GM of SARS-CoV-2 neutralizing titers in all participants | At D01 and D30
  SARS-CoV-2 neutralizing titers
GMR of SARS-CoV-2 neutralizing titers ratio D30/D01 in all participants | At D01 and D30
  Individual SARS-CoV-2 neutralizing titers ratio D30/D01

SECONDARY OUTCOMES:
Percentage of participants with seroconversion in all participants | At D30
  Seroconversion is defined by:
  HAI titer < 10 [1/dil] at D01 and post-injection titer ≥ 40 [1/dil] at D30 or HAI titer ≥ 10 [1/dil] and a ≥ 4-fold increase in titer [1/dil] at D30
Percentage of participants with HAI titer ≥ 10 (1/dil) in all participants | At D01 and D30
  detectable HAI titer ≥ 10 (1/dil)
Percentage of participants with HAI titer ≥ 40 (1/dil) in all participants | At D01 and D30
  HAI titer ≥ 40 (1/dil)
Percentage of participants with seroresponse to SARS-CoV-2 in all participants | At D30
  Seroresponse to SARS-CoV-2 is defined by SARS-CoV-2 neutralizing titers ≥ 4-fold rise in SARS-CoV-2 neutralizing titers from D01 to D30

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Simon Williamson Clinic - Birmingham- Site Number : 8400003, Birmingham, Alabama
  - AES - DRS - Optimal Research Alabama - Huntsville Site Number : 8400006, Huntsville, Alabama
  - Orange Grove Family Practice- Site Number : 8400012, Tucson, Arizona
  - Synexus Clinical Research US, Inc. - The Villages Site Number : 8400011, The Villages, Florida
  - Synexus Clinical Research US - Atlanta- Site Number : 8400001, Atlanta, Georgia
  - Synexus Clinical Research- Site Number : 8400004, Chicago, Illinois
  - Synexus Clinical Research - St. Louis- Site Number : 8400010, Creve Coeur, Missouri
  - Synexus New York Site Number : 8400007, New York, New York
  - Optimal Research, LLC Site Number : 8400002, Austin, Texas
  - Synexus Clinical Research US - Dallas- Site Number : 8400005, Dallas, Texas
  - Synexus Clinical Research US - San Antonio- Site Number : 8400009, San Antonio, Texas
  - Synexus Salt Lake City Site Number : 8400008, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org